CLINICAL TRIAL: NCT02935803
Title: A Prospective and Randomised Single Centre Study on the Anti-incontinent Effectiveness of the Modified Trans Vaginal Mesh Method in POPQ Stage II-III Patients
Brief Title: A Study on the Anti-incontinent Effectiveness of the mTVM Method in POPQ Stage II-III Patients
Acronym: TVMvsmTVM
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Szeged University (Other)
Responsible Party: Principal Investigator, Zoltan Fekete, assistant lecturer, Szeged University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: TVM/mTVM 55/2016
Record Dates: First submitted 2016-05-20; First posted 2016-10-18 (Estimated); Last update posted 2016-10-18 (Estimated); Status verified 2016-10

CONDITIONS: Uterine Prolapse; Urinary Stress Incontinence; Side Effects
MeSH Terms: conditions — Uterine Prolapse; Urinary Incontinence, Stress

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Modified TVM operation (Other): Modified Trans-vaginal Mesh operation (mTVM): polypropylene monofilament meshes produced by Aspide® fixed up to the mid urethra by a resolvable suture. 76 participants will be involved.
  Interventions: Procedure: Trans-vaginal Mesh operation
- Control group (Other): 76 Participants as control group undergo a traditional Trans-vaginal Mesh operation (TVM) with polypropylene monofilament meshes produced by Aspide® . (Sergent et al.)
  Interventions: Procedure: Trans-vaginal Mesh operation

INTERVENTIONS:
Procedure: Trans-vaginal Mesh operation — Modified the transobturator TVM operation reported by Sergent et al. by inserting a stabilizing suture, which fixing the anterior edge of the mesh to the paraurethral tissues at the level of the mid-urethra with two non-resolvable anchoring stitches thereby promoting the proper elevation and closure of the urethra

SUMMARY:
An increasing number of specific procedures have been described for the surgical repair of pelvic organ prolapse (POP) and concomitant stress urinary incontinence (SUI). The investigators introduced an alternative operative method for POP-Q II-III repair and anti-incontinence with the trans vaginal mesh (TVM) anterior edge fixed to the periurethral tissues at the level of mid-urethra. The efficacy and short- and long-term complication profile, of this new surgical technique as compared with those of non-modified TVM.

DETAILED DESCRIPTION:
The prospective randomized double blind study comprised 152 women who presented for the correction of stress urinary incontinence (SUI) in conjunction with anterior compartment pelvic organ prolapse stage II-III (POP-Q II-III) at the Departments of Obstetrics and Gynecology at the University of Szeged, Hungary, between June of 2016 and June 2017. After a block randomization method, the patients will divide into two arms, the study group which consist of 76 patients will undergo modified trans vaginal mesh operation (TVM), the rest 76 patients as a control group will undergo a traditional TVM operation. Inclusion criteria in the study is coexisting SUI and POP Q St II-III and signature of the informed consent. The exclusion criteria are as follows: urge, mixed or neurogenic incontinence, occult SUI, previous mesh operations, anti-depressive medical therapy, cancer of the pelvic organs, urinary infections, any sign of voiding difficulties. The transobturator TVM operation (Sergent et al.) has been modofied by inserting a stabilizing suture, which fixing the anterior edge of the mesh to the para-urethral tissues at the level of the mid-urethra with two non-resolvable anchoring stitches thereby promoting the proper elevation and closure of the urethra. The hypothesis is the stabilizing suture treat the coexisting SUI as well. In all cases, urodynamic examinations were carried out before the surgery and urodynamic examinations comprising uroflowmetry, cystography and Valsalva leak point pressure tests and pelvic floor ultrasonography will be performed to determine the coexisting SUI. The efficacy of the POP repair is taken as a significant (>1 cm) improvement at points Aa, Ba, C and D according to the POP-Q system (International Continence Society) during the follow-up. The anti-incontinence efficacy is classified as no further SUI diagnosed by urodynamic examination and pelvic floor sonography. All patients will fill two validated Hungarian language questionnaires as "A short form of the Pelvic Organ Prolapse/Urinary Incontinence Sexual Questionnaire" (PISQ-12) and "Pelvic Floor Distress Inventory" PFDI. After a one-year application phase all patients will be followed for 36 months. During follow- up phase repeated urodynamic studies, pelvic floor sonography urine culturing will be done after 3, 12, 24 and 36 months. The evaluation of the POP-Q system and Bonney's cough test and the PISQ-12 and PFDI questionnaires will be performed at every regular check-ups

ELIGIBILITY:
Inclusion Criteria:

* Coexisting SUI and POP Q St II-III and signature of the informed consent

Exclusion Criteria:

* Urge, mixed or neurogenic incontinency, occult SUI, previous mesh operations, antidepressive medical therapy, cancer of the pelvic organs, urinary infections, any sign of voiding difficulties

Ages: 45 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 76 (Estimated)
Dates: Start 2016-07; Primary Completion 2017-06 (Estimated); Study Completion 2020-06 (Estimated)

PRIMARY OUTCOMES:
Efficacy of the mTVM on genuine stress incontinence. | 36 months flollow up
  Measuring the anti incontinence effect of the used method by urodynamic examination anf pelvic floor sonography

SECONDARY OUTCOMES:
Telorability of the mTVM method | 36 month follow up
  Measuring the tolerability of the used method by the Clavien-Dindo classification system
Improvement in sexual life | 36 month
  Define the change in quality of sexual life after the used procedures by Pelvic Organ Prolapse/Urinary Incontinence Sexual Questionnaire (PISQ-12)
Improvement in pelvic floor symphtoms | 3 years follow up
  Define the change in quality of life after the used procedures by Pelvic Floor Distress Inventory (PFDI-20)
Improvement in quality of life | 3 years
  Define the change in quality of life after the used procedures by urogenital distress inventory (UDI-6)

CONTACTS AND LOCATIONS:
Overall Officials: Zoltan Fekete, M.D., Principal Investigator — Szeged University; Gábor Németh, M.D., Ph.D., Study Director — Szeged University
Locations (1):
- Univ. of Szeged. Dep. of Obstetrics and Gynaecology, Szeged, Hungary

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Background] Minassian VA, Stewart WF, Wood GC. Urinary incontinence in women: variation in prevalence estimates and risk factors. Obstet Gynecol. 2008 Feb;111(2 Pt 1):324-31. doi: 10.1097/01.AOG.0000267220.48987.17. PMID 18238969
- [Background] Kirss F, Lang K, Toompere K, Veerus P. Prevalence and risk factors of urinary incontinence among Estonian postmenopausal women. Springerplus. 2013 Oct 17;2:524. doi: 10.1186/2193-1801-2-524. eCollection 2013. PMID 24171152
- [Background] Akkus Y, Pinar G. Evaluation of the prevalence, type, severity, and risk factors of urinary incontinence and its impact on quality of life among women in Turkey. Int Urogynecol J. 2016 Jun;27(6):887-93. doi: 10.1007/s00192-015-2904-5. Epub 2015 Dec 5. PMID 26638154
- [Background] Tinelli A, Malvasi A, Rahimi S, Negro R, Vergara D, Martignago R, Pellegrino M, Cavallotti C. Age-related pelvic floor modifications and prolapse risk factors in postmenopausal women. Menopause. 2010 Jan-Feb;17(1):204-12. doi: 10.1097/gme.0b013e3181b0c2ae. PMID 19629013
- [Background] Molander U, Milsom I, Ekelund P, Mellstrom D. An epidemiological study of urinary incontinence and related urogenital symptoms in elderly women. Maturitas. 1990 Apr;12(1):51-60. doi: 10.1016/0378-5122(90)90060-j. PMID 2333037
- [Background] Lau HH, Huang WC, Cheng YW, Wang H, Su TH. Changes in urodynamic measurements and bladder neck position after single-incision trans-vaginal mesh for pelvic organ prolapse. Int Urogynecol J. 2015 Nov;26(11):1629-35. doi: 10.1007/s00192-015-2753-2. Epub 2015 Jul 10. PMID 26156205
- [Background] Sergent F, Gay-Crosier G, Bisson V, Resch B, Verspyck E, Marpeau L. Ineffectiveness of associating a suburethral tape to a transobturator mesh for cystocele correction on concomitant stress urinary incontinence. Urology. 2009 Oct;74(4):765-70. doi: 10.1016/j.urology.2009.05.038. Epub 2009 Jul 30. PMID 19643459
- [Derived] Fekete Z, Suranyi A, Renes L, Nemeth G, Kozinszky Z. Efficacy of anchoring the four-arm transvaginal mesh to the mid-urethra vs original surgery as a surgical correction for stress urine incontinence in coexisting anterior vaginal prolapse grades II and III: study protocol for a randomized controlled trial. Trials. 2017 Dec 28;18(1):624. doi: 10.1186/s13063-017-2314-8. PMID 29282115
- See also: Surge-Mesh Prolapse by Aspide is used for both TVM method — http://www.aspide.com/en/gynecological-urological-surgery/p/surgimesh-prolapse